CLINICAL TRIAL: NCT06708624
Title: An Open-Label, Multi-Center, Single-Arm Study to Evaluate the Ocular Safety and Usability of FYB201 Pre-filled Syringe (PFS)
Brief Title: Ocular Safety and Usability Study for FYB201 PFS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Formycon AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FYB201-C3-02
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Age-Related Macular Degeneration; Branch Retinal Vein Occlusion with Macular Edema; Central Retinal Vein Occlusion with Macular Edema
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FYB201 0.5 mg (0.05 mL of 10 mg/mL) (Experimental): FYB201 provided in a pre-filled syringe (PFS), containing 0.5 mg of 10 mg/mL ranibizumab in 0.05 mL for intravitreal (IVT) administration
  Interventions: Drug: FYB201 0.5 mg (0.05 mL of 10 mg/mL)

INTERVENTIONS:
Drug: FYB201 0.5 mg (0.05 mL of 10 mg/mL) — IVT administration of FYB201 in a PFS
  Other Names: ranibizumab-eqrn

SUMMARY:
The objective of the study is to assess the ocular safety of the FYB201 pre-filled syringe in terms of preparation and administration by Retina Specialists in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

1. Study eye deemed to be indicated for ranibizumab intravitreal injection therapy at the discretion of the Investigator.
2. Written and signed informed consent form (ICF) obtained before any study-related procedures are performed.
3. Have a confirmed diagnosis in one or both eyes of Neovascular (Wet) Age-Related Macular Degeneration (AMD) or Macular Edema Following Retinal Vein Occlusion (RVO).
4. Qualifies for treatment with ranibizumab-eqrn according to the USPI.
5. Aged ≥18 years at the time of signing ICF.
6. If a subject is already on a ranibizumab regimen, timing of study participation should correlate with the regimen.
7. Male study subject (if his female spouse/partner is of childbearing potential) must confirm that he is using two acceptable methods for contraception (one of which must be a barrier method) starting at signing ICF and throughout the clinical study period and for 3 months after study drug administration. Male study subject should agree to inform his partner of participation in the study and the need to avoid pregnancy. Surgically sterilized and non-sexually active male subjects do not require additional use of contraception.
8. Male study subject agrees not to donate sperm starting from screening and throughout the clinical study period and for 3 months after study drug administration.
9. Female study subject must be categorized by at least one of the following:

   * Not a Woman of Child-bearing Potential as described in Appendix 3 prior to signing ICF; or
   * Surgically sterile or having undergone a hysterectomy as categorized in Appendix 3 at least 1 month prior to signing ICF; or
   * Is using a highly effective contraception. All females of childbearing potential will be required to use highly effective contraception (as described in Appendix 3) starting at signing ICF and throughout the clinical study period and for 3 months after study drug administration.
10. Female study subject must not be lactating and must not be breastfeeding at screening until 3 months after study drug administration.
11. Female study subject must not donate ova starting at signing ICF and throughout the clinical study period and for 3 months after study drug administration.

Exclusion Criteria:

1. Have received IVT injection in the study eye within 3 months prior to Day 1 with any anti-VEGF therapy other than ranibizumab products (e.g. Lucentis®, Cimerli®, Byooviz®).
2. Intraocular corticosteroid administration in the study eye within 30 day prior to Day 1.
3. The study subject has/had fever or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to Day 1.
4. The study subjects with a history or evidence of SARS-CoV-2 infection in the last month prior to signing ICF or having been in confirmed contact with SARS-CoV-2 positive patients in the last 2 weeks before dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Incidence and occurrence of ocular and non-ocular Adverse Events (AEs) and Serious Adverse Events (SAEs) occurring after IVT injection | 2 days
  To assess the ocular safety of the FYB201 PFS in terms of preparation and administration by Retina Specialists.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Site, Campbell, California
  - Research Site, Long Beach, California
  - Research Site, Hagerstown, Maryland
  - Research Site, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: No